CLINICAL TRIAL: NCT06516185
Title: Randomized Clinical Trial on the Efficacy and Effectiveness of Two Types of Aligners Based on Stratification by Type of Movement.
Brief Title: Efficacy and Effectiveness of Two Types of Aligners Based on Stratification by Type of Movement
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 125-120324; 24/098-EC_P (Registry Identifier: Ethics Committee for Research involving medicinal products (IECm))
Record Dates: First submitted 2024-07-08; First posted 2024-07-23 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-06

CONDITIONS: Crowding, Tooth; Tipped Tooth or Teeth; Rotation of Tooth; Malocclusion, Angle's Class
Keywords: clear aligner therapy; direct-printed aligner; predictability; shape memory; stratification
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Intervention Model Description: This study is designed following CONSORT guidelines as a randomized equivalence clinical trial, controlled, with two parallel arms, and single-blind.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct-printed aligner (Experimental): The experimental group will be treated with the aligner system fabricated by direct printing. The current protocols described in the literature and by the manufacturer for the fabrication of the printed orthodontic devices will be followed.
  Interventions: Device: direct-printed aligner
- Thermoformed aligner (Active Comparator): The control group will be treated with the thermoformed or gold standard aligner system. The established protocols for treatment with thermoformed clear aligners will be followed.
  Interventions: Device: thermoformed aligner

INTERVENTIONS:
Device: direct-printed aligner — Patients will be treated with direct-printed aligners until dental alignment is achieved.
  Arms: Direct-printed aligner
Device: thermoformed aligner — Patients will be treated with thermoformed aligners until dental alignment is achieved.
  Arms: Thermoformed aligner

SUMMARY:
The purpose of this study is to evaluate the biomechanical behaviour of direct-printed and thermoformed aligners in different tooth movements, creating a biomechanical planning protocol based on a stratification of tooth movements according to the degree of predictability.

DETAILED DESCRIPTION:
Once the objectives, benefits, risks and follow-up of the study have been explained to each eligible patient, patients will be asked to sign an informed consent form. They will also be informed that they may cancel their participation in the study at any time. Patient will be allocated randomly in two groups: The first group will receive orthodontic treatment with direct-printed aligner, while the second group will receive orthodontic treatment with conventional or gold standard thermoformed aligner.

ELIGIBILITY:
Inclusion Criteria:

* Patients with malocclusion and invididual dental malpositions requiring orthodontic treatment
* Adequate oral and periodontal health, with absence of periodontal disease, periapical infection or untreated caries.
* No history of previous orthodontic treatment.
* Complete permanent dentition (excluding third molars, their presence or absence being irrelevant).

Exclusion Criteria:

* Altered bone metabolism (including use of antiresorptive, steroid or immunosuppressive drugs).
* Pregnant women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Predictability for each type of tooth movement in patients with direct-printed aligners compared to a control group in which the movements are performed with thermoformed aligners. | Baseline and when the defined endpoint (crowding resolution, LII=0) is reached, an average of six months.
  The primary outcome will be quantified through a continuous numerical variable, tooth movement efficiency or predictability (%) measured as the change between the final, intra-treatment and initial position for each of the individual movements studied, expressed as a percentage (%). The end of treatment or endpoint (E1) of this study will be established when the measurement of Little's Irregularity Index (hereafter LII) LII=0.
impact on the effectiveness and predictability of biomechanics auxiliaries compared to a control group in which movements are performed without the use of auxiliaries. | Baseline and when the defined endpoint (crowding resolution, LII=0) is reached, an average of six months.
  This will be assessed by quantifying the change between the predictability with auxiliaries and without auxiliaries for each of the individual movements studied respectively, expressed as a percentage (%).

SECONDARY OUTCOMES:
PROMs of the patient undergoing direct-printed aligner treatment compared to the control group. | These should be completed five times after each visit (at 24 hours, 48 hours, 72 hours, 7 days and 14 days of aligner use) until reaching the defined endpoint (crowding resolution, LII=0), an average of 6 months.
  Participants will complete a validated pre-defined questionnaire [Patient-reported outcome measures (PROMs)] on treatment use and perceptions. The level of pain will be assessed using questionnaires.
influence on the printed orthodontic device (POD) of varying the degree of inclination of the aligner print. | Baseline and when the defined endpoint (crowding resolution, LII=0) is reached, an average of six months.
  This will be assessed by quantifying the change between the predictability, varying the degree of inclination of the aligner print, expressed as a percentage (%).

CONTACTS AND LOCATIONS:
Locations (1):
- Complutense University of Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available at the end of the clinical trial in June 2026
Access Criteria: Upon request of the interested party